CLINICAL TRIAL: NCT01224691
Title: The Role of TGF-Beta in Asthmatic Epithelial Cell Susceptibility to RSV Infection
Brief Title: TGF-(Beta) and Susceptibility to RSV
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110006; 11-E-0006
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-08-14

CONDITIONS: Asthma
Keywords: TGF-Beta; Asthma; Natural History; Healthy Volunteer; Respiratory Syncytial Virus; RSV
MeSH Terms: conditions — Asthma; Camurati-Engelmann Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asmathics: Asmathics
- Non-Asmathics: Non-Asmathics

SUMMARY:
Background:

* Human respiratory syncytial virus (RSV) is a virus that causes respiratory tract infections, and is frequently responsible for hospital visits in infants and children. It can also trigger severe breathing problems for individuals who have asthma, but these infections are generally better tolerated in non-asthmatics. Some research suggests that lack of an efficient immune system response in people with asthma may make it difficult for the body to fight the effects of RSV.
* Transforming Growth Factor-beta (TGF-[beta]) is a chemical in the body that is more prevalent in the lungs of people with asthma and related respiratory disorders. More information is needed about the effects of TGF-[beta] and whether it makes individuals with asthma more prone to developing RSV. Researchers hope to use this information to determine possible treatments and therapies for individuals with asthma who contract RSV.

Objectives:

- To determine the possible role of TGF-[beta] in increased asthmatic susceptibility to RSV infection.

Eligibility:

- Individuals between 18 and 60 years of age who are either healthy nonsmokers or mild asthmatics.

Design:

* This study involves a screening visit and a study visit.
* Participants will be screened with a medical history and physical examination, as well as blood samples and a pulmonary function test.
* At the study visit, participants will receive mild anesthetic and have a bronchoscopy, in which researchers insert a bronchoscope through the participant s nose or mouth and into the lungs to examine the lungs and collect lung cells.
* Participants will be contacted by a research team member 24 36 hours after the bronchoscopy to ask about any side effects from the procedure.

DETAILED DESCRIPTION:
This is a cross-sectional, controlled study designed to investigate whether Transforming Growth Factor-beta (TGF-beta) mediates increased asthmatic epithelial susceptibility to respiratory syncytial virus (RSV) infection by examining responses to RSV infection in epithelial cells cultured from asthmatic and non-asthmatic participants. Non-smoking healthy adults and mild asthmatics, aged 18-60 years old, will be recruited to participate. Potential participants will be prescreened and scheduled for a final eligibility visit that will include medical history review, vital signs, physical examination, blood draw, and pulmonary function tests (PFTs). After eligibility is confirmed, the participant will be scheduled for bronchoscopy. During the bronchoscopy, bronchial epithelia and alveolar macrophages will be obtained from the participant for analysis. Alveolar macrophages will be evaluated ex-vivo for inflammatory activity at baseline and after stimulation.

The primary objective of the laboratory analysis is to determine if TGF-beta mediates increased asthmatic epithelial susceptibility to RSV infection. The study has three aims which are interrelated: 1) To determine if asthmatic bronchial epithelia express more TGF-beta than normal epithelia; 2) to determine if RSV replication is greater in asthmatic epithelia than normal epithelia; and 3) to determine if TGF-beta mediates asthmatic bronchial epithelial susceptibility to RSV infections.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Male or female between 18 and 60 years of age
2. Non-asthmatics and mild asthmatics as defined below:

   * Non-asthmatic must have no prior diagnosis of asthma, no history of health care utilization or medication use for asthma, no current symptoms, and Forced Expiratory Volume in 1 Second (FEV1) greater than or equal to 80% predicted.
   * Asthmatics must have physician-diagnosed asthma for at least one year and evidence of mild, persistent disease during the month prior to Visit 1 (based on 2008 GINA guidelines).

     a) Participants who are currently taking a controller medication must:

     i. use the equivalent to GINA Step 1 or 2 therapy; and

   ii. have controlled disease, as defined by:
   * daytime symptoms less than or equal to 2 times week, such as wheezing, tightness in the chest, shortness of breath, and cough,
   * no nocturnal symptoms;

     b) Participants who are not currently taking a controller must have:

     i.<TAB>daytime symptoms > 1 time a week but < 1 time a day, such as wheezing, tightness in the chest, shortness of breath, and cough;

   ii. nocturnal awakenings > 2 times a month but < 1 time a week;

   c) All asthmatic participants must have either:

   i.<TAB>Pre-bronchdilator FEV1 greater than or equal to 80% predicted and a positive methacholine challenge (PC20 less than or equal to 4 mg / ml); or

   ii.<TAB>Pre-bronchodilator FEV1 < 80% and post-bronchodilator FEV1 greater than or equal to 80% with significant bronchodilator reversibility (at least 12% or 200ml change in FEV1)
3. Participants must be able to understand and provide written informed consent
4. Participants must be able to travel to the CRU and the EPA

EXCLUSION CRITERIA:

1. Use of oral steroid treatment(s) within 30 days of Visit 1
2. Acute asthma-related healthcare utilization within 30 days of Visit 1, such as ED visits, systemic corticosteroids, and nebulizer treatment for asthma exacerbation
3. Known or suspected respiratory infections within 30 days of Visit 1, such as flu, pneumonia, severe cold, tuberculosis, or bronchitis
4. Known or suspected viral infection within 30 days of Visit 1
5. History of chronic obstructive pulmonary disease other than asthma
6. History of immunological disease or current cancer
7. Uncontrolled cardiovascular disease such as angina, prior myocardial infarction, stroke, and high cholesterol
8. Cardiac malformations
9. Pulmonary hypertension
10. Bleeding disorders
11. Facial deformity, major facial surgery
12. Currently pregnant or breast feeding
13. Current smoker, significant second-hand smoke exposure (defined by urine cotinine > 100 ng/ml at Visit 1 or Visit 2) or former smokers (defined by a history of smoking > 100 cigarettes)
14. Insulin dependent diabetes
15. Used any of the following medications within 30 days of Visit 1: oral corticosteroids, systemic immunosuppressants or other immune-modifying drugs [e.g., Rituxan, Humira, Enbrel, Azathioprine (Imuran), Cyclosporine (Neoral, Sandimmune, and SangCya), cyclophosphamide, TNF antagonists], anticoagulants (clopidogrel, heparin, enoxaparin and related drugs, coumadin), and sustained use (i.e. more than one dose per day for more than two days) of non-steroidal anti-inflammatory drugs (aspirin, ibuprofen, indomethacin) within seven days of bronchoscopy
16. Allergy or history of adverse reactions to methacholine or lidocaine
17. Severe asthma as defined by a history of intubation for unstable asthma
18. Any condition that, in the investigator's opinion, places the participant at undue risk for complications (e.g. from PFTs, fiberoptic bronchoscopy, bronchalveolar lavage and/or bronchial brushings)
19. Temperature > 37.6 C; blood pressure < 90/50 mm Hg or blood pressure >170/95 mm Hg; pulse rate < 50 or > 100 beats/minute
20. Body weight < 50 kg (<110 lbs)
21. The following abnormal lab values (values obtained during clinical assessment):

    * Platelet count < 100,000 per 10(9)/L
    * White blood cells count < 3000 per 10(9)/L
    * Hematocrit < 35% for both female and male
    * Prothrombin Time (PT) / Abnormal International Normalized Ratio (INR) and partial prothromboplastin time (PTT) based on reference laboratory established reference ranges
    * Serum creatinine > 1.4 mg/dL

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be individuals from the Research Triangle Park (RTP) area in North Carolina (see Section 6.2.1 for Recruitment Methods). Participants will be between the ages of 18 and 60 years and will be 1) healthy non-asthmatics and 2) mild asthmatics defined by 2008 Global Initiative for Asthma (GINA) criteria.@@@
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2012-03-19 (Actual)

PRIMARY OUTCOMES:
The primary hypothesis for Aim 1 is that asthmatics: cultured epithelia will have higher TGF-Beta expression levels than non-asthmatics. | analysis
  If En and Ea are the means of the logarithms of expression levels for the normal (non-asthmatic) and asthmatic populations, respectively, then the null hypothesis is H1,0: En = Ea and the one-sided alternative hypothesis is H1,0: En < Ea. This hypothesis will be tested with a one-sided, two-sample t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Garantziotis, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
It has not been decided yet if we will share the data

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-E-0006.html